CLINICAL TRIAL: NCT02613858
Title: Minimal HePatic Encephalopathy Among CiRrhotics. A Cross SEctional, Clinico-EpidEmiological, Multi-Centre, Study in Patients of PakisTan
Acronym: Preempt
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Dimension Research (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIDI038
Record Dates: First submitted 2015-11-06; First posted 2015-11-25 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Preempt study is likely to help determine the frequency of patients suffering from Minimal Hepatic Encephalopathy (MHE) and are cirrhotics. It will also enable us to know about the Quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex, 18-65 years of age, who have attended school at least till the 5th Class/Standard having an established diagnosis of liver cirrhosis without any overt symptoms at time of testing with Grade 0 of West Haven criteria.
* Patients willing to undergo the neuropsychological (NP) tests and to complete the SF-36 questionnaire for the estimation of Health Related Quality of Life (HRQOL).
* Patients willing to provide written authorization to provide data for the study.

Exclusion Criteria:

* Patients with inability to perform neuropsychometric tests and to complete the SF-36 questionnaire as decided by the physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic/Private Clinic
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Frequency of MHE in Cirrhotic patients | 18 months
  Continuous variables with normal and non-normal distributions would be reported as mean (SD) and median [inter-quartile range (IQR)], respectively. Prevalence of MHE in cirrhotic patients with 95% confidence Interval (CI) will be calculated. Continuous variables between group will compared by using Independent sample t test, and categorical variables will compare by using the chi-square test.

SECONDARY OUTCOMES:
The predisposing factors that might be associated with MHE in all enrolled patients with cirrhosis | 18 months
  Odds Ratios (OR) and their 95% Confidence Intervals (CI) will be estimated using Logistic Regression. The likelihood ratio test used to assess the association between the explanatory variables and the risk of the MHE. Invariable analyses will perform to examine the effect of each variable on the risk of MHE. In multivariate analysis all insignificant variables (p >0.05) will check for their confounding and interaction effects before their removal from the final model.
Quality of Life (QoL) of patients at baselines | 18 months
  Short Form (SF)-36v2 Quality of Life Questionnaire will be used
Management of MHE currently in practice | 18 months
  As per practice of the physician/Investigator. Management of MHE will be recorded. The information for medication which will be collected will be Name (preferably the generic name), Dose, Units (form of the medicine), Route and Frequency

CONTACTS AND LOCATIONS:
Overall Officials: Raeefuddin Ahmed, MD, Study Director — Medical Director, Abbott
Locations (6):
- Pakistan (6):
  - Baqai Hospital, Karachi
  - Fatima Memorial Hospital, Lahore
  - Lahore General Hospital, Lahore
  - Jinnah Hospital Lahore, Lahore
  - Doctor's Hospital, Lahore
  - Lady Reading Hospital, Peshawar